CLINICAL TRIAL: NCT04563429
Title: Vitamin A Oral Supplementation as a Preventive Treatment for Chronic Lung Disease Among Infants Born Before 29 Weeks of Gestation.
Brief Title: Vitamin A for BPD Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Leah Leibovitch MD, MD, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SHEBA-20-7281-LL-CTIL
Record Dates: First submitted 2020-09-22; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: The Relationship Between Oral Vitamin A Administration and the Incidence of BPD in Preterm Infants Born Before Week 29 of Pregnancy
MeSH Terms: interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Dietary Supplement: Oral Vitamin A
- Control Group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Oral Vitamin A — Oral administration of 5000 EU of Vitamin A during first 28 days of life
  Arms: Treatment Group

SUMMARY:
Chronic bronchopulmonary dysplasia (BPD) is a very common complication in preterm infants born at a young gestational age, and is a serious disease that impairs respiratory long-term outcome and is associated with higher-frequency neurodevelopmental injury. Lowering the incidence of BPD may improve the health of the preterm babies and neurodevelopmental delay of preterm infants.Vitamin A deficiency may be one of the factors associated with the development of BPD in preterm infants. According to the literature, oral vitamin A administration can lower the incidence of BPD. In our study we plan to give 5000 units of retinol / dose / day, every day for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Premature babies under 29 weeks, at any birth weight
* A preterm baby is less than 4 days to life

Exclusion Criteria:

* Major congenital malformations
* Known chromosomal disorders

Ages: 2 Days to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of BPD at 28 days | 28 days of life
  Chronic pulmonary desease of prematue babies
Incidence of mortality at 28 days | 28 days of life
  Death before 28 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Leah Leibovich, MD, Principal Investigator — Chaim Sheba Medical Center, Tel Hashomer, Israel

IPD SHARING:
Plan to Share IPD: No